CLINICAL TRIAL: NCT02904928
Title: Incidence and Perioperative Factors Associated With Postoperative Delirium Among Surgical Patients in Mulago National Referral Hospital
Brief Title: Incidence and Perioperative Factors Associated With Postoperative Delirium
Acronym: iPOD
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/HDO7/611
Record Dates: First submitted 2016-08-04; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With the increasing number of advanced surgical operations being done annually, including the elderly, the risk of developing postoperative delirium is potentially high. Postoperative delirium is associated with longer hospital stay, poorer functional outcome, cognitive decline and an elevated morbidity and mortality, in addition to an increased cost of health care. However, most of the studies on postoperative delirium have been done in high income countries, leaving a paucity of literature on the incidence and associated factors of postoperative delirium in Africa and hence a need to do this study.

DETAILED DESCRIPTION:
The paucity of literature in the low income setting as regards to the complication of post operative delirium has led to under recognition and under diagnosis of this problem.The lack of diagnostic tools, such as the CAM, has contributed to low rates of diagnosis and index of suspicion among clinicians.

Objectives were To determine the incidence and perioperative factors associated with postoperative delirium in adult patients undergoing elective surgery in Mulago National Referral Hospital (MNRH) Procedure Patient recruitment Patients were stratified by ward and then systematic sampling was used with a sampling interval of 3. On each day of recruitment, the first 3 patients on the theatre list on a particular ward were selected by writing numbers 1 to 3 on pieces of paper and randomly selecting one; the number selected would be the first to be enrolled, succeeded by every 3rd patient on the theatre list for that day. Written informed consent was obtained preoperatively from each study patient.

Preoperative assessment Trained research assistants conducted the preoperative interviews with a questionnaire within 12 hours before surgery. Patient demographics, pain scores, Glasgow coma scores, smoking history, alcohol consumption, anaesthetic history, American Society of Anaesthesiologists (ASA), Class as recorded on the anaesthetic chart, vitals and laboratory results of complete blood count, renal and liver functional tests available were recorded.

Delirium assessment To determine the presence of delirium, research assistants conducted structured interviews preoperatively and on the first three postoperative days between hours of 9am and 12 pm, using the Confusion Assessment Method (CAM). Based on a structured interview, the CAM algorithm included four clinical criteria: acute onset and fluctuating course, inattention, disorganized thinking, and altered level of consciousness. To define delirium, both the first and second criteria had to have been present, plus either criterion three or four. The research assistants were trained in CAM use.

To ensure consistency in the evaluation, each patient was evaluated by the same research assistant for all three interviews. All cases of incident delirium were validated by a second investigator. The investigators focused on delirium measurement on the first 3 days postoperatively, aiming to avoid loss to follow up as the majority of postoperative patients in our setting get discharged on the third postoperative day.

Associated factors Risk factors identified during the preoperative interviews included age, history of smoking and alcohol use, preoperative pain scores, medications, and electrolytes. Other factors including type of surgery, ASA classification, duration of anaesthesia, Intraoperative blood loss as recorded on the anaesthetic charts. Blood loss was estimated using the common method of adding up volumes of blood absorbed in the commonly used absorptive materials including the gauze pieces, sponges and the mops. Suction canisters measured pre and post operatively and calculated minus the irrigation used in the case. Then the total estimated intraoperative blood loss was charted on the anaesthetic chart, intraoperative medications were obtained from the anaesthetic chart.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients above 18 years who have consented to participate in the study and are fully conscious by the Glasgow coma scale

Exclusion Criteria:

* Patients with psychiatric disease confirmed by medical documents, as these were unable to provide informed consent
* Patients undergoing neuro surgery and open heart surgery, as these patients were expected to remain intubated postoperatively, precluding cognitive assessments.
* Patients scheduled for emergency surgery. Sample size Estimation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with surgical disease admitted on the surgical wards in Mulago National Referral Hospital scheduled for surgery during the study period who met the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative delirium | 72 hours
  the CAM assessment tool was administered preoperative and then delirium assessed postoperatively at the times given above using a CAM diagnostic tool administered by research assistant.when the patient was CAM positive at any time they were discontinued from the study

SECONDARY OUTCOMES:
perioperative factors associated with postoperative delirium | up to 72 hours
  using a pretested questionnaire, perioperative factors were assessed

CONTACTS AND LOCATIONS:
Overall Officials: JOSHUA SEMPIIRA, MBCHB, Principal Investigator — MAKERERE UNIVERSITY DEPARTMENT OF ANAETHESIA; DICKENS H AKENA, PHD, Study Director — MAKERERE UNIVERSITY DEPARTMENT OF PSYCHIATRY; EMMANUEL T AYEBALE, MMED, Study Director — MAKERERE UNIVERSITY DEPARTMENT OF ANAESTHESIA; AGNES WABULE, MMED, Study Chair — MAKERERE UNIVERSITY DEPARTMENT OF ANAESTHESIA
Locations (1):
- Mulago Hospital Complex, Kampala, Kampala, Uganda